CLINICAL TRIAL: NCT05211661
Title: Development of Diaphragm Atrophy, Dysfunction and Inhibited Cortical Control in Mechanical Ventilation
Brief Title: Diaphragm Atrophy and Dysfunction in Mechanical Ventilation
Acronym: DAM
Status: Recruiting | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Principal Investigator, Univ.-Prof. Dr. med. Michael Dreher, Professor Michael Dreher, RWTH Aachen University
Other Study IDs: CTCA 21-279
Record Dates: First submitted 2022-01-04; First posted 2022-01-27 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Diaphragm Issues; Mechanical Ventilation Complication; Respiratory Failure; Intensive Care (ICU) Myopathy
MeSH Terms: conditions — Respiratory Insufficiency; Muscular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples obtained based on venous puncture
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Invasively ventilated patients (n=15): First measurement (comprehensive protocol) within 48 hours from initiation of MV.
  Serial measurements every third day including 2 measurements after extubation.
  Interventions: Diagnostic Test: Respiratory Muscle Testing

INTERVENTIONS:
Diagnostic Test: Respiratory Muscle Testing — Comprehensive assessment of respiratory muscle function. Comprehensive assessment of respiratory muscle function to the point of its invasive assessment with recordings of twitch transdiaphragmatic pressure in response to magnetic phrenic nerve stimulation and stimulation of the lower thoracic nerve roots.

SUMMARY:
The gold standard of twitch transdiaphragmatic pressure recordings would ultimately clear the fog around the rate of development of Ventilator induced Diaphragm Dysfunction (VIDD) in mechanically ventilated patients over time.

Through measurements made even after mechanical ventilation (MV) it could be clarified to what extent patients recover from VIDD.

Paired with cortical stimulation and electromyographic recordings of diaphragm muscle potentials, it could be explored to what extent decreased diaphragm excitability due to long term MV contributes to VIDD on the level of motor cortex.

Against that background the present project aims at determining the rate of decline in diaphragm function, strength and control in patients undergoing MV (including measurements after extubation).

DETAILED DESCRIPTION:
Evidence both from animal and human studies support the development of ventilator induced diaphragm dysfunction (VIDD) from as early as 24 hours of mechanical ventilation (MV) in the intensive care unit (ICU).

However, while the concept of VIDD seems to be proven now, several questions remain unanswered regarding its actual rate of development and (potentially) recovery after MV.

The gold standard of twitch transdiaphragmatic pressure recordings would ultimately clear the fog around the rate of development of VIDD over time.

Through measurements made even after MV it could be clarified to what extent patients recover from VIDD.

Paired with cortical stimulation and electromyographic recordings of diaphragm muscle potentials, it could be explored to what extent decreased diaphragm excitability due to long term MV contributes to VIDD on the level of motor cortex.

Against that background the present project aims at determining the rate of decline in diaphragm function, strength and control in patients undergoing MV (including measurements after extubation).

ELIGIBILITY:
Inclusion Criteria:

* Initiation of invasive mechanical ventilation in the Intensive Care Unit within 48 hours.
* Expected duration of invasive mechanical ventilation of at least 5 days.

Exclusion Criteria:

* Body-mass-index (BMI) >40
* Expected absence of active participation of the patient in study-related measurements after extubation
* Alcohol or drug abuse
* Non MRI compatible implant in the body
* Slipped disc
* Epilepsy
* Patients in an interdependence or with an employment contract with the principal investigator, Co-PI or his deputy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Comprehensive assessment of diaphragm atrophy, function, strength and control in patients in whom invasive mechanical ventilation in the Intensive Care Unit had been initiated within 48 hours. Then, serial measurements every third day including 2 measurements after extubation.
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Twitch transdiaphragmatic pressure in response to supramaximal magnetic stimulation of the phrenic nerve roots. | 2 years
Cortical control of diaphragm function | 2 years
  Amplitude of the diaphragm motor evoked potentials (measured by surface electrodes attached to the diaphragm) following cortical magnetic stimulation of the phrenic nerve roots.

SECONDARY OUTCOMES:
Diaphragm ultrasound | 2 years
  Diaphragm thickening fraction on ultrasound
Systemic inflammation | 2 years
  Concentration of circulating Interleukin, high-sensitivity C-reactive protein (analyzed quantitatively based on a Levels venous blood sample).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dreher, Professor, Study Chair — RWTH Aachen University Hospital; Jens Spiesshoefer, MD, Principal Investigator — RWTH Aachen University Hospital
Locations (1):
- RWTH Aachen University, Aachen, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Spiesshoefer J, Herkenrath S, Henke C, Langenbruch L, Schneppe M, Randerath W, Young P, Brix T, Boentert M. Evaluation of Respiratory Muscle Strength and Diaphragm Ultrasound: Normative Values, Theoretical Considerations, and Practical Recommendations. Respiration. 2020;99(5):369-381. doi: 10.1159/000506016. Epub 2020 May 12. PMID 32396905
- [Background] Spiesshoefer J, Henke C, Herkenrath S, Randerath W, Brix T, Young P, Boentert M. Assessment of Central Drive to the Diaphragm by Twitch Interpolation: Normal Values, Theoretical Considerations, and Future Directions. Respiration. 2019;98(4):283-293. doi: 10.1159/000500726. Epub 2019 Jul 26. PMID 31352459
- [Background] Spiesshoefer J, Henke C, Herkenrath S, Brix T, Randerath W, Young P, Boentert M. Transdiapragmatic pressure and contractile properties of the diaphragm following magnetic stimulation. Respir Physiol Neurobiol. 2019 Aug;266:47-53. doi: 10.1016/j.resp.2019.04.011. Epub 2019 Apr 25. PMID 31029769
- [Background] Sharshar T, Ross ET, Hopkinson NS, Porcher R, Nickol AH, Jonville S, Dayer MJ, Hart N, Moxham J, Lofaso F, Polkey MI. Depression of diaphragm motor cortex excitability during mechanical ventilation. J Appl Physiol (1985). 2004 Jul;97(1):3-10. doi: 10.1152/japplphysiol.01099.2003. Epub 2004 Mar 12. PMID 15020575
- [Background] Windisch W, Geiseler J, Simon K, Walterspacher S, Dreher M; on behalf of the Guideline Commission. German National Guideline for Treating Chronic Respiratory Failure with Invasive and Non-Invasive Ventilation: Revised Edition 2017 - Part 1. Respiration. 2018;96(1):66-97. doi: 10.1159/000488001. Epub 2018 Jun 26. PMID 29945148
- [Background] Windisch W, Geiseler J, Simon K, Walterspacher S, Dreher M; on behalf of the Guideline Commission. German National Guideline for Treating Chronic Respiratory Failure with Invasive and Non-Invasive Ventilation - Revised Edition 2017: Part 2. Respiration. 2018;96(2):171-203. doi: 10.1159/000488667. Epub 2018 Jun 26. PMID 29945156